CLINICAL TRIAL: NCT04415229
Title: Seasonality of Respiratory Syncytial Virus (RSV) Bronchiolitis in Children Aged 2 Years or Less Hospitalized in Martinique (French West Indies) a Tropical Area From 2007 to 2018
Brief Title: RSV Seasonality in Martinique in Children Aged 2 Years or Less
Acronym: VRS-12
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 19_MR004-11
Record Dates: First submitted 2020-04-09; First posted 2020-06-04 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Bronchiolitis; Respiratory Syncytial Virus
Keywords: Bronchiolitis; Respiratory Syncytial Virus; Child; Infant, premature; Bronchopulmonary Dysplasia; Heart Defects, Congenital; Tropical climate; Humidity; Epidemiology; Air pollution
MeSH Terms: conditions — Bronchiolitis; Premature Birth; Bronchopulmonary Dysplasia; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The epidemiological characteristics of RSV bronchiolitis differ between tropical and temperate zones. This study seeks to understand which climatic factors could influence the specific seasonality of these bronchiolitis in Martinique and to verify the hypothesis put forward: influence of favorable climatic conditions in the month preceding the start of the epidemic. In addition, the study will improve our knowledge of the epidemiology of the infection in order to improve the management of infants.

DETAILED DESCRIPTION:
Respiratory Syncytial Virus (RSV) infections are the leading cause of hospitalization for respiratory distress in infants (50% of children under 1 year of age are infected with the virus, 100% of children under 3 years of age). They are responsible for 66,000 to 199,000 deaths in children under 5 years of age worldwide, and 15,000 to 20,000 hospitalizations in France depending on the year. It is a highly contagious virus whose transmission is both respiratory and by hand and which appreciates humidity to develop.

In temperate regions where this infection has been well studied, it occurs preferentially during the winter, probably favoured by the cold and humidity, as well as by the confinement of individuals during this season. The more the child is young, premature, has a chronic respiratory pathology or congenital heart disease, the more sever the disease. Prevention is based on the injection of a monoclonal antibody (Palivizumab) before the start of the epidemic season and on conventional hygiene measures. But today, little epidemiological data is available for tropical regions and in Martinique, which makes it impossible to understand why, how and when RSV develops on our island. Some epidemiological studies carried out in tropical regions point to the possibility that the humidity in the air would favour viral development and in fact, these epidemics are more frequently found during the rainy season. The humidity level, the number of rainy days, the rate of sunshine and cloud cover, and finally the importance of the wind, could explain a different seasonality from that known in temperate regions (seasonality being linked to the virus circulation patterns and being defined as the ability to re-emerge at the same period from one year to the next).

Research issues A first study carried out at the University hospital of Martinique over a period of 2 years (from July 1, 2007 to December 31, 2008) has made it possible to specify the epidemiology a little better but the results need to be confirmed. This work seems to show that the epidemic starts earlier than in temperate zones: (late August - early September to late November - early December) versus (November - December to March - April) respectively. The number of cases per epidemic can change significantly (factor 2.5). However, this first study was not long enough to ensure that the seasonality identified will be systematically repeated from one year to the next. Moreover, this study did not allow us to specify the number of children with clinical severity criteria on our island.

By carrying out a study over a longer period, the investigators will have a better understanding of seasonality and the rate of disease in children in Martinique, allowing us to better anticipate the extent and severity of these phenomena. This precision will allow us to determine when to start Monoclonal Antibody injections for vulnerable children (essentially infants with chronic respiratory pathologies or congenital cardiac pathologies, i.e. approximately 30 children per year in Martinique). The investigators will also be able to anticipate future needs of beds and caregivers to the epidemic to come or in progress. The investigators will therefore have better preventive care for children at risk and better preparation of the healthcare offer.

Research questions

* Descriptions of the characteristics of RSV bronchiolitis epidemics (seasonality, rate of occurrence, case profile)?
* What are the factors that may explain a specific seasonality and case rate in tropical zones, especially Martinique? What is the role of climatic factors?

Research hypotheses The investigators believe that the seasonality and characteristics of RSV bronchiolitis are indeed specific to tropical areas such as Martinique.

The investigators hypothesize that, in tropical areas, certain favourable climatic conditions, prevailing in the month prior to the usual period of RSV bronchiolitis outbreak onset or during the epidemic, would be intrinsically linked to the characteristics of these epidemics.

Indeed, RSV is a virus that particularly likes humid atmospheres in which to develop. These conditions are conducive during the rainy season in the tropics (second half of the year in Martinique), which could explain a different seasonality from that known in temperate regions (where the epidemic occurs rather during the winter). These favourable climatic conditions can be approximated by measuring the humidity level, the number of rainy days, the average temperature, the rate of sunshine and cloud cover and the average wind strength. In addition, respiratory irritants such as sand mist or other air pollution, as assessed by the air quality index, could be among the parameters that explain these differences.

The investigators propose to retrospectively analyze 12 years of hospital data on RSV bronchiolitis cases in Martinique among hospitalized children 2 years of age and younger, the main targets of RSV, and therefore the population most vulnerable to this virus. The investigators will focus only on hospitalized patients because they are the most severely affected patients, which will allow us to accurately describe the clinical severity criteria in this at-risk population.

Main objective Describe the temporal distribution of RSV bronchiolitis cases in children 2 years of age or younger hospitalized in Martinique, over a 12-year period (2007 to 2018), based on climatic parameters prevailing in the month before the beginning of the epidemic or during the epidemic.

Secondary objectives

* Describe the weekly and monthly distribution of RSV bronchiolitis, over the 12-year study period, among children 2 years of age and younger hospitalized in Martinique.
* Describe the characteristics of each epidemic observed over the study period.
* Describe the characteristics of RSV bronchiolitis cases during the study period.
* Analyze the association between the climatic parameters studied and the occurrence of RSV bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* two years of age or younger
* hospitalized for bronchiolitis in the pediatrics department of the University hospital of Martinique over the period 2007 to 2018
* with a confirmed virological diagnosis of RSV virus by ImmunoFluorescence (IF) from 01/01/2007 to 31/01/2016 and from 01/02/2016 by Reverse transcription polymerase chain reaction.
* with a clinical diagnosis of bronchiolitis (presentation of suggestive clinical signs such as cough, respiratory distress associated with a febrile illness, with rhinopharyngitis in the previous days)
* no opposition from the legal representative for the use of the data from the medical file in the context of the research. This non-opposition is documented in the patient's medical file

Exclusion Criteria:

* opposition from the legal representative for the use of the data from the medical file
* Inability to inform legal representatives of the conduct of the research

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children 2 years of age or younger hospitalized in Martinique with RSV bronchiolitis cases, over a 12-year period (2007 to 2018)
Sampling Method: Probability Sample
Enrollment: 1237 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Incident cases of RSV bronchiolitis in children between 2007 and 2018 | 1 year
  Monthly distribution of incident cases of RSV bronchiolitis in children aged 2 years or less hospitalized from 2007 to 2018 (number of cases/month) according to the values of the following climatic parameters recorded during the month preceding the beginning of the epidemic or during the epidemic : 7-day average humidity (%)
Incident cases of RSV bronchiolitis in children between 2007 and 2018 | 1 year
  Monthly distribution of incident cases of RSV bronchiolitis in children aged 2 years or less hospitalized from 2007 to 2018 (number of cases/month) according to the values of the following climatic parameters recorded during the month preceding the beginning of the epidemic or during the epidemic : number of significant rainy days (j)
Incident cases of RSV bronchiolitis in children between 2007 and 2018 | Through study completion, an average of 1 year
  Monthly distribution of incident cases of RSV bronchiolitis in children aged 2 years or less hospitalized from 2007 to 2018 (number of cases/month) according to the values of the following climatic parameters recorded during the month preceding the beginning of the epidemic or during the epidemic : average temperature (°C) over one day
Incident cases of RSV bronchiolitis in children between 2007 and 2018 | 1 year
  Monthly distribution of incident cases of RSV bronchiolitis in children aged 2 years or less hospitalized from 2007 to 2018 (number of cases/month) according to the values of the following climatic parameters recorded during the month preceding the beginning of the epidemic or during the epidemic : global solar radiation (joules/cm²)
Incident cases of RSV bronchiolitis in children between 2007 and 2018 | 1 year
  Monthly distribution of incident cases of RSV bronchiolitis in children aged 2 years or less hospitalized from 2007 to 2018 (number of cases/month) according to the values of the following climatic parameters recorded during the month preceding the beginning of the epidemic or during the epidemic : average wind force (km/h)
Incident cases of RSV bronchiolitis in children between 2007 and 2018 | 1 year
  Monthly distribution of incident cases of RSV bronchiolitis in children aged 2 years or less hospitalized from 2007 to 2018 (number of cases/month) according to the values of the following climatic parameters recorded during the month preceding the beginning of the epidemic or during the epidemic : concentrations, in µg/m3, of air pollutants (such as nitrogen oxides (NOx) and fine particulate matter (PM10))
RSV cases by month compare with climatic factors at the same time | Through study completion, an average of 1 year
  Climatic parameters: 7-day average humidity (%)
RSV cases by month compare with climatic factors at the same time | 1 year
  Climatic parameters: number of significant rainy days (j)
RSV cases by month compare with climatic factors at the same time | 1 year
  Climatic parameters: average temperature (°C) over one day
RSV cases by month compare with climatic factors at the same time | 1 year
  Climatic parameters: solar radiation (joules/cm²)
RSV cases by month compare with climatic factors at the same time | 1 year
  Climatic parameters: average wind force (km/h)
RSV cases by month compare with climatic factors at the same time | 1 year
  Climatic parameters: concentrations, in µg/m3, of air pollutants such as nitrogen oxides (NOx) and fine particulate matter (PM10).

SECONDARY OUTCOMES:
Distribution of RSV bronchiolitis | 1 year
  Weekly and monthly distribution of RSV bronchiolitis
Distribution of RSV bronchiolitis | By week
  Weekly distribution of RSV bronchiolitis
Distribution of RSV bronchiolitis | Through study completion, an average of 1 year
  Monthly distribution of RSV bronchiolitis
Characteristics of each epidemic | 1 year
  Characteristics of each epidemic (beginning, peak and end of epidemic; number of incident cases per week, month and year; incidence curve per week, month and year; rate of attainment (cumulative incidence of infection over the period))
Characteristics of incident cases | 1 year
  Characteristics of incident cases: sex, age, hospitalization in pediatric ICU, oxygen therapy, assisted respiration rate, enteral nutrition rate, prematurity, chronic respiratory pathology of the former prematurity, congenital heart disease.)
Climatic parameters and RSV bronchiolitis | 1 year
  Correlation between the climatic parameters studied and the occurrence of RSV bronchiolitis

CONTACTS AND LOCATIONS:
Overall Officials: Olivier FLECHELLES, MD, Principal Investigator — Hospital University of Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bont L, Checchia PA, Fauroux B, Figueras-Aloy J, Manzoni P, Paes B, Simoes EA, Carbonell-Estrany X. Defining the Epidemiology and Burden of Severe Respiratory Syncytial Virus Infection Among Infants and Children in Western Countries. Infect Dis Ther. 2016 Sep;5(3):271-98. doi: 10.1007/s40121-016-0123-0. Epub 2016 Aug 1. PMID 27480325
- [Background] RAMEIX-WELTI M, GAULT E. Le virus respiratoire syncytial (VRS): état actuel des connaissances. Feuill. Biol. 2017;29-41.
- [Background] Welliver TP, Garofalo RP, Hosakote Y, Hintz KH, Avendano L, Sanchez K, Velozo L, Jafri H, Chavez-Bueno S, Ogra PL, McKinney L, Reed JL, Welliver RC Sr. Severe human lower respiratory tract illness caused by respiratory syncytial virus and influenza virus is characterized by the absence of pulmonary cytotoxic lymphocyte responses. J Infect Dis. 2007 Apr 15;195(8):1126-36. doi: 10.1086/512615. Epub 2007 Mar 9. PMID 17357048
- [Background] Paes B, Fauroux B, Figueras-Aloy J, Bont L, Checchia PA, Simoes EA, Manzoni P, Carbonell-Estrany X. Defining the Risk and Associated Morbidity and Mortality of Severe Respiratory Syncytial Virus Infection Among Infants with Chronic Lung Disease. Infect Dis Ther. 2016 Dec;5(4):453-471. doi: 10.1007/s40121-016-0137-7. Epub 2016 Nov 18. PMID 27864751
- [Background] Checchia PA, Paes B, Bont L, Manzoni P, Simoes EA, Fauroux B, Figueras-Aloy J, Carbonell-Estrany X. Defining the Risk and Associated Morbidity and Mortality of Severe Respiratory Syncytial Virus Infection Among Infants with Congenital Heart Disease. Infect Dis Ther. 2017 Mar;6(1):37-56. doi: 10.1007/s40121-016-0142-x. Epub 2017 Jan 9. PMID 28070870
- [Background] Sande CJ, Mutunga MN, Medley GF, Cane PA, Nokes DJ. Group- and genotype-specific neutralizing antibody responses against respiratory syncytial virus in infants and young children with severe pneumonia. J Infect Dis. 2013 Feb 1;207(3):489-92. doi: 10.1093/infdis/jis700. Epub 2012 Nov 21. PMID 23175761
- [Background] Yamaguchi M, Sano Y, Dapat IC, Saito R, Suzuki Y, Kumaki A, Shobugawa Y, Dapat C, Uchiyama M, Suzuki H. High frequency of repeated infections due to emerging genotypes of human respiratory syncytial viruses among children during eight successive epidemic seasons in Japan. J Clin Microbiol. 2011 Mar;49(3):1034-40. doi: 10.1128/JCM.02132-10. Epub 2010 Dec 22. PMID 21177891
- [Background] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- [Result] Equipe de surveillance de la bronchiolite. Surveillance de la bronchiolite en France, saison 2016-2017. Bull Epidémiol Hebd. 2017;650-657.